CLINICAL TRIAL: NCT03006406
Title: Effect of Shorten Gonadotropin-releasing Hormone Agonist Therapy on the Outcome of in Vitro Fertilization-Embryo Transfer in Patients With Endometriosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yingpu Sun, Director of Reproductive Medical Center,1st Affilated Hospital, Zhengzhou University, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO-1
Record Dates: First submitted 2016-12-28; First posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Clinical Pregnancy Rate
Keywords: endometriosis; long term GnRH-a
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Long term GnRH-a for 1 month (Active Comparator): patient in this group only receive GnRH-a 3.75 for 1 month
  Interventions: Drug: Long term GnRH-a (3.75mg)
- patient in this group only receive GnRH-a 3.75 for 2 month (Experimental): patient in this group only receive GnRH-a 3.75 for 2 month
  Interventions: Drug: Long term GnRH-a (3.75mg)

INTERVENTIONS:
Drug: Long term GnRH-a (3.75mg) — patient in this group only receive GnRH-a 3.75 for pituitary down-regulation

SUMMARY:
Gonadotropin-releasing hormone analogue (GnRH-a) is a synthetic decapeptide compound which can down-regulate pituitary function causing a temporary low estrogen state. Since endometriosis is an estrogen-dependent disease, the use of long-acting GnRH-a can control the growth of endometriosis by inhibiting ovary function.Some scholars have found that, for adenomyosis patients who received a super long protocol (pretreatment of long-acting GnRH-a for 1-2 months) in IVF treatment, the pregnancy outcome is comparable to that of the controls with normal uterus. Thus, the aim of this study is to compare the clinical pregnancy rate in patients treated with GnRH-a for 1, or 2 months.

ELIGIBILITY:
Inclusion Criteria:

* first IVF cycle;
* with normal ovarian reserve(FSH(10miu/ml； antral follicle count )3)
* with normal uterine

Exclusion Criteria:

* Pre-implantation genetic diagnosis cycles;
* Oocyte donation cycles

Ages: 22 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 5 weeks after embryo transfer

SECONDARY OUTCOMES:
Number of oocytes retrieved | 1 day at oocyte retrieved day
2 pronucleus(2PN)fertilization rate | 48hours after oocyte retrieved day
  Number of 2PN/Matured oocytes

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medical Center, First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van der Houwen LE, Mijatovic V, Leemhuis E, Schats R, Heymans MW, Lambalk CB, Hompes PG. Efficacy and safety of IVF/ICSI in patients with severe endometriosis after long-term pituitary down-regulation. Reprod Biomed Online. 2014 Jan;28(1):39-46. doi: 10.1016/j.rbmo.2013.09.027. Epub 2013 Oct 9. PMID 24262434
- [Background] Mijatovic V, Florijn E, Halim N, Schats R, Hompes P. Adenomyosis has no adverse effects on IVF/ICSI outcomes in women with endometriosis treated with long-term pituitary down-regulation before IVF/ICSI. Eur J Obstet Gynecol Reprod Biol. 2010 Jul;151(1):62-5. doi: 10.1016/j.ejogrb.2010.02.047. Epub 2010 Apr 21. PMID 20409633
- [Derived] Kong H, Hu L, Nie L, Yu X, Dai W, Li J, Chen C, Bu Z, Shi H, Wu Q, Guan Y, Sun Y. A multi-center, randomized controlled clinical trial of the application of a shortened protocol of long-acting Triptorelin down-regulated prior to IVF/ICSI among patients with endometriosis: A protocol. Reprod Health. 2018 Dec 20;15(1):213. doi: 10.1186/s12978-018-0639-8. PMID 30572916